CLINICAL TRIAL: NCT00994474
Title: Comparison of Clinical Outcome Parameters, the Patient Benefit Index (PBI) and Patient Satisfaction After Ablative Fractional Laser Treatment of Peri-orbital Rhytides
Brief Title: Comparison of Outcome Parameters in Laser Rhytide Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laserklinik Karlsruhe (Other)
Responsible Party: Christian Raulin/Professor Dr., Laserklinik Karlsruhe
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: LK_06_2009
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Skin Aging
Keywords: Laser surgery; Profilometry; Fitzpatrick wrinkle score; Patient Benefit Index; Patient satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fractional carbon dioxide laser treatment (Active Comparator)
  Interventions: Procedure: Fractional carbon dioxide laser treatment
- Fractional Er:YAG laser treatment (Active Comparator)
  Interventions: Procedure: Fractional Er:YAG laser treatment

INTERVENTIONS:
Procedure: Fractional carbon dioxide laser treatment — With the CO2 laser (Fraxel Re:pair, Solta Medical Inc., Hayward, CA), patients received two passes at 15 mJ (1st pass) and 20 mJ (2nd pass), respectively, with a total density of 20 %. We employed 'pin-point bleeding' and serosanguinous exudate as a clinical end point. The pulse duration was 10 msec.
  Arms: Fractional carbon dioxide laser treatment
Procedure: Fractional Er:YAG laser treatment — The Er:YAG laser (MCL 30 Dermablate, Asclepion Laser Technologies GmbH, Jena, Germany) was used in 4 passes with a total fluence of 60 J/cm² and pulse stacking (6 stacked pulses); the pulse duration was 400 μsec.
  Arms: Fractional Er:YAG laser treatment

SUMMARY:
We previously published a comparative split-face study which has shown a significant, albeit moderate, effect of ablative fractional laser treatment. While indicating that a single session with fractional ablative lasers can be effective in the treatment of peri-orbital wrinkles, the trial also revealed substantial disagreement between the different end points (profilometry, Fitzpatrick wrinkle score, patient satisfaction). Since the PBI is a patient-related index it could not be included in the aforementioned split-face trial; the present study therefore attempts to further elucidate the patient-related benefit of a single fractional ablative laser treatment session as well as carefully analyse the respective correlations between the outcome parameters employed.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate peri-orbital rhytides ('crow's feet') at rest (Class II according to Fitzpatrick)

Exclusion Criteria:

* unrealistic expectations
* inability to meet follow-up criteria
* Fitzpatrick skin phototype >III
* coagulation disorders or anti-coagulant treatment
* allergy to lidocaine or tetracaine
* oral isotretinoin within the last 6 months
* any active skin disease within the treatment areas (e.g., psoriasis, cancer, or autoimmune disease)
* synthetic implants in the treatment area
* facial cosmetic procedures affecting the treatment area within the last 6 months
* photosensitizing medications (e.g., tetracycline, gold)
* history of keloid formation
* pregnancy

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2008-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Quantitative measurement of wrinkle depth | Before and after treatment (3 months)
Fitzpatrick wrinkle score | Before and after treatment (3 months)

SECONDARY OUTCOMES:
Patient benefit index (PBI) | Before and after treatment (3 months)
Patient satisfaction | 1, 3, 6 days and 3 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Syrus Karsai, MD, Principal Investigator — Laserklinik Karlsruhe
Locations (1):
- Laserklinik Karlsruhe, Karlsruhe, Germany